CLINICAL TRIAL: NCT02615821
Title: Mental Contrasting Physical Activity Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: H14-02120
Record Dates: First submitted 2015-11-19; First posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Exercise; Attitude to Health; Motivation; Goals
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Affective Mental Contrasting (Experimental): Before the goal formation or mental contrasting activities, participants will receive information about the affective benefits of exercising (e.g. regular physical activity has been shown to reduce stress, physical activity is enjoyable), and related research support including appropriate references. During the mental contrasting component of the activity the prompts will remain the same as the standard condition, with minor variations in questions in order to elicit affective judgements. Specifically, the affective condition will include the additional prompts "Why might you find exercise to be enjoyable, pleasant, exciting, or fun?" for eliciting outcomes, and "Why might you find exercise to be unenjoyable, unpleasant, boring, or miserable?" for eliciting obstacles.
  Interventions: Behavioral: Mental Contrasting
- Instrumental Mental Contrasting (Active Comparator): Before the goal formation or mental contrasting activities,participants will receive information about the instrumental benefits of exercising (e.g., regular physical activity reduces the risk of developing cancer) and related research support, again including appropriate references. During the mental contrasting component of the activity the prompts will remain the same as the standard condition, with minor variations in questions in order to elicit either instrumental judgements. Specifically, the instrumental conditions will include the prompts "Why might you find exercise to be useful, advantageous, beneficial, or important?" for eliciting outcomes, and "Why might you find exercise to be unimportant, useless, inconvenient, or detrimental?" for eliciting obstacles.
  Interventions: Behavioral: Mental Contrasting
- Standard Mental Contrasting (Active Comparator): In the standard condition, the space where the affective and instrumental benefits of physical activity were listed in the instrumental and affective conditions, will be left blank in the standard condition, and no additional prompting questions will be given, allowing for the idiosyncratic identification of obstacles and outcome.
  Interventions: Behavioral: Mental Contrasting

INTERVENTIONS:
Behavioral: Mental Contrasting — n the mental contrasting activity participants will be asked by the researcher to consider the best outcome associated with engaging in physical activity, as well as the obstacles they may encounter while completing the activity. The first question will ask participants to name the most positive outcome of realizing their goal (e.g., feeling more awake during classes; weight loss). The second question will ask participants to name the most critical obstacle (e.g., feeling tired; rain) to reaching their goal.

SUMMARY:
Given the numerous physical and psychological benefits of engaging in regular physical activity (Biddle & Ekkekakis, 2005; Warburton et al., 2007) and the decrease in students' physical activity levels during the transition from high school to university (Bray & Born, 2010) it is important for researchers to develop time-and-cost-effective interventions to prevent this drop in physical activity. Intervention research shows mental contrasting (a goal setting strategy) can be taught in a cost-and-time-effective way in order to increase physical activity (Oettingen, 2012). Researchers have also found that individuals who consider the emotional effects of physical activity are more likely to be physically active than those who consider the health-related effects (Rhodes et al., 2009). The purpose of this research is to combine these two approaches to develop and evaluate a novel mental contrasting intervention to increase physical activity among a sample of undergraduate students.

DETAILED DESCRIPTION:
The transition from high school to university is a vulnerable period for discontinuing regular physical activity, which can have implications for individuals' physical and psychological health (Bray & Born, 2010). Accordingly, it is imperative to find and implement cost and time-effective interventions to mitigate the consequences of this transition. Mental contrasting is a goal-setting strategy that involves imagining the greatest outcome associated with achievement of a desired future goal while considering the aspects of one's present situation that may serve as obstacles for attaining that same goal (Oettingen & Gollwitzer, 2010). Intervention research has shown that mental contrasting can be taught as a metacognitive strategy in a cost- and time-effective way, affecting numerous health behaviours including physical activity (Oettingen, 2012). Drawing from diverse theoretical perspectives (e.g., Bechara, 2005; Lawton, Conner, & McEachan, 2009; Williams, 2010), recent meta-analytic evidence suggests that affective judgements (e.g., enjoyable-unenjoyable) exert greater influence on physical activity behaviors than health-related instrumental judgements (e.g., useful-useless; Rhodes, Fiala, & Conner, 2009). Nevertheless, research has yet to utilize mental contrasting as a means of targeting affective judgements, through intervention, in order to bolster physical activity promotion efforts. This research will examine how an affective mental contrasting intervention will change university students' affective judgements in comparison to instrumental mental contrasting and standard mental contrasting comparison conditions, and the subsequent impact of these changes on physical activity behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Individuals will be eligible to participate if they are female, inactive (i.e., engage in moderate-vigorous intensity physical activity for more than 30 minutes, less than three times a week), studying for an undergraduate degree at the University of British Columbia, and are able to read and converse in English.

Exclusion Criteria:

* Participants will be excluded if they have any self-reported physical health conditions using the online version of the PAR-Q+ (http://eparmedx.com/?page_id=75) that would restrict them from increasing their physical activity behaviours at the time of the intervention.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change is accelerometry measured moderate-vigorous physical activity from baseline | One week immediately following the intervention
  Actigraph accelerometers will measure daily activities. A standard 7-day accelerometry monitoring protocol will be used. Participants will also complete three one-week physical activity logs corresponding to the three accelerometry periods. In these logs, participants will record the time the monitor is on and off, in addition to recording all activities performed with or without the monitor.
Change is accelerometry measured moderate-vigorous physical activity from baseline | Four-week follow-up
  Actigraph accelerometers will measure daily activities. A standard 7-day accelerometry monitoring protocol will be used. Participants will also complete three one-week physical activity logs corresponding to the three accelerometry periods. In these logs, participants will record the time the monitor is on and off, in addition to recording all activities performed with or without the monitor.

SECONDARY OUTCOMES:
Change in Godin's Leisure Time Exercise Questionnaire (GLTEQ) | Change between baseline and four-week follow-up
  Participants will report the typical number of minutes per week they engaged in mild, moderate, and vigorous physical activity. As per the protocol for scoring the GLTEQ, physical activity is transformed into MET hours by multiplying hours of engagement in mild physical activity by 2, moderate activity by 4, and vigorous physical activity by 7, and then summing these values to provide an estimate of MET hours/week for each of the two time points assessed.
Change is Affective and Instrumental Physical Activity Judgements | Changes between baseline, the week immediately following the intervention, and a four-week follow-up.
  Instrumental and affective judgements towards participants' physical activity goal will be measured using semantic differential scales (Ajzen, 2002). Five items will be used to tap instrumental judgements (e.g. 'For me, engaging in moderate to vigorous aerobic physical activity for at least 150 minutes a week for the next 6 weeks would be': useless-useful), and five items will be used to tap affective judgements (e.g. 'For me, engaging in moderate to vigorous aerobic physical activity for at least 150 minutes a week for the next 6 weeks would be': unenjoyable-enjoyable). Each adjective pair will be rated on a 7-point unipolar scale (1-7) and a mean score will be computed for instrumental and affective subscales respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Beauchamp, Principal Investigator — University of British Columbia
Locations (1):
- Psychology of Exercise, Health, and Physical Activity Laboratory, University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Ruissen GR, Rhodes RE, Crocker PRE, Beauchamp MR. Affective mental contrasting to enhance physical activity: A randomized controlled trial. Health Psychol. 2018 Jan;37(1):51-60. doi: 10.1037/hea0000551. Epub 2017 Oct 5. PMID 28981303